CLINICAL TRIAL: NCT05984251
Title: A Double-blind, Placebo-controlled, Single and Multiple Ascending Dose Phase 1 Study to Evaluate the Safety, Tolerability, and Pharmacokinetics of CCX168 in Healthy Male and Female Subjects
Brief Title: A Study to Evaluate the Safety, Tolerability, and Pharmacokinetics of CCX168 in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Basic Science
Other Study IDs: CL001_168
Record Dates: First submitted 2023-08-02; First posted 2023-08-09 (Actual); Last update posted 2023-08-09 (Actual); Status verified 2023-08

CONDITIONS: Vasculitis; Systemic Lupus Erythematosus (SLE)
Keywords: Complement; C5aR; Vascular diseases; Cardiovascular diseases
MeSH Terms: conditions — Vasculitis; Lupus Erythematosus, Systemic; Vascular Diseases; Cardiovascular Diseases | interventions — avacopan

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Cohort 1 (Experimental): During Period 1, participants will receive a single dose of CCX168 1 mg or placebo. During the second study period, participants will receive the same dose as during the first period but once daily (QD) for a period of 7 days continuously.
  Interventions: Drug: CCX168; Drug: Placebo
- Cohort 2 (Experimental): During Period 1, participants will receive a single dose of CCX168 3 mg or placebo. During the second study period, participants will receive the same dose as during the first period but QD for a period of 7 days continuously.
  Interventions: Drug: CCX168; Drug: Placebo
- Cohort 3 (Experimental): During Period 1, participants will receive a single dose of CCX168 10 mg or placebo. During the second study period, participants will receive the same dose as during the first period but QD for a period of 7 days continuously.
  Interventions: Drug: CCX168; Drug: Placebo
- Cohort 4 (Experimental): During Period 1, participants will receive a single dose of CCX168 30 mg or placebo. During the second study period, participants will receive the same dose as during the first period or placebo twice daily (BID) for a period of 7 days continuously.
  Interventions: Drug: CCX168; Drug: Placebo
- Cohort 5 (Experimental): During Period 1, participants will receive a single dose of CCX168 100 mg or placebo. During the second study period, participants will receive the same dose as during the first period or placebo BID for a period of 7 days continuously.
  Interventions: Drug: CCX168; Drug: Placebo

INTERVENTIONS:
Drug: CCX168 — Administered orally.
Drug: Placebo — Administered orally.

SUMMARY:
The primary objective of this study will be to evaluate the safety and tolerability of single and multiple oral doses of CCX168, over a range of dose levels, in healthy male and female participants.

ELIGIBILITY:
Inclusion Criteria:

* Male or female participants, aged 19-45 years inclusive, who are in generally good health, whose body mass index is 19 to 29 kg/m^2;
* Willing and able to give written Informed Consent and to comply with the requirements of the study protocol;
* Negative result of the human immunodeficiency virus screen, the hepatitis B screen, and the hepatitis C screen;
* Judged to be healthy by the Investigator, based on medical history, physical examination (including ECG), and clinical laboratory assessments. Participants with clinical laboratory values that are outside of normal limits and/or with other abnormal clinical findings that are judged by the Investigator not to be of clinical significance may be entered into the study, and
* Female participants of childbearing potential, and male participants with partners of childbearing potential, may participate if adequate contraception is used during, and for at least the four weeks after, any administration of study medication.

Exclusion Criteria:

* Women who are pregnant, breastfeeding, or have a positive serum pregnancy test at Screening and/or on Study Day -1;
* Expected requirement for use of any medication (with the exception of continuing use by female participants of hormonal contraceptives in accordance with a regimen that has been stable for at least the three months prior to Screening) during the study period;
* History within the three months prior to study entry of use of tobacco and/or nicotine containing products;
* History within one year prior to study entry of illicit drug use;
* History of alcohol abuse at any time in the past;
* History of any form of cancer;
* Consumed alcoholic beverages, or any food or drink containing grapefruit or grapefruit juice within 24 hours of screening;
* History or presence of any medical condition or disease which, in the opinion of the Investigator, may place the participant at unacceptable risk for study participation;
* Donated or lost more than 350 mL of blood or blood products within 56 days prior to Screening, or donated plasma within 7 days of randomization;
* Participant's hemoglobin less than 12 g/dL (or less than 7.45 mmol/L);
* Participated in any clinical study of an investigational product within 30 days prior to randomization;
* Participant has any evidence of hepatic disease; aspartate aminotransferase, alanine aminotransferase, gamma-glutamyl transpeptidase, alkaline phosphatase, or bilirubin > 1.5 x the upper limit of normal;
* Participant has any evidence of renal impairment; serum creatinine > 1.5 x upper limit of normal, and
* Participant's urine tested positive at Screening and/or on Study Day -1 for any of the following: opioids, amphetamines, cannabinoids, benzodiazepines, barbiturates, cocaine, cotinine, or alcohol (Breathalyzer test allowed for alcohol).

Ages: 19 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2009-12-21 (Actual); Primary Completion 2010-09-19 (Actual); Study Completion 2011-04-11 (Actual)

PRIMARY OUTCOMES:
Number of Participants Experiencing Adverse Events (AEs) | Up to 43 days
Number of Participants Experiencing Clinically Significant Changes in Laboratory Parameters | Up to 29 days
Number of Participants Experiencing Clinically Significant Changes in Electrocardiogram (ECG) Parameters | Up to 29 days
Number of Participants Experiencing Clinically Significant Changes in Vital Sign Parameters | Up to 29 days

SECONDARY OUTCOMES:
Maximum Plasma Concentration (Cmax) of CCX168 | Period 1: Up to Day 8; Period 2: Up to Day 15
Time of Cmax of CCX168 | Period 1: Up to Day 8; Period 2: Up to Day 15
Terminal Phase Rate Constant of CCX168 | Period 1: Up to Day 8; Period 2: Up to Day 15
Apparent Terminal Half-life of CCX168 | Period 1: Up to Day 8; Period 2: Up to Day 15
Apparent Oral Clearance of CCX168 | Period 1: Up to Day 8; Period 2: Up to Day 15
Apparent Volume of Distribution of CCX168 | Period 1: Up to Day 8; Period 2: Up to Day 15
Area Under the Plasma Concentration-time Curve (AUC) of CCX168 From Time 0 to Time t | Period 1: Up to Day 8; Period 2: Up to Day 15
AUC of CCX168 From Time 0 to Infinity | Period 1: Up to Day 8; Period 2: Up to Day 15
AUC of CCX168 From Time 0 to 24 Hours | Periods 1 and 2: Up to Hour 24
AUC of CCX168 From Time 0 to 12 Hours | Periods 1 and 2: Up to Hour 12
AUC of CCX168 From Time 12 to 24 Hours | Periods 1 and 2: Hour 12 to Hour 24
Period 2: AUC of CCX168 From Time 0 to the end of the Dosing Interval | Cohorts 1-3: Up to Hour 24; Cohorts 4-5: Up to Hour 12
Period 2: Accumulation Ratio of CCX168 | Up to Day 7
Percent Inhibition of complement 5a receptor (C5aR)-dependent Upregulation of CD11b in Peripheral Blood Neutrophils | Period 1: Up to Hour 24; Period 2: Up to 12 hours after the first dose on Day 7

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (1):
- Covance Clinical Research Unit (CRU) AG, Allschwil, Switzerland

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual patient data for variables necessary to address the specific research question in an approved data sharing request.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data sharing requests relating to this study will be considered beginning 18 months after the study has ended and either 1) the product and indication have been granted marketing authorization in both the US and Europe or 2) clinical development for the product and/or indication discontinues and the data will not be submitted to regulatory authorities. There is no end date for eligibility to submit a data sharing request for this study.
Access Criteria: Qualified researchers may submit a request containing the research objectives, the Amgen product(s) and Amgen study/studies in scope, endpoints/outcomes of interest, statistical analysis plan, data requirements, publication plan, and qualifications of the researcher(s). In general, Amgen does not grant external requests for individual patient data for the purpose of re-evaluating safety and efficacy issues already addressed in the product labelling. Requests are reviewed by a committee of internal advisors. If not approved, a Data Sharing Independent Review Panel will arbitrate and make the final decision. Upon approval, information necessary to address the research question will be provided under the terms of a data sharing agreement. This may include anonymized individual patient data and/or available supporting documents, containing fragments of analysis code where provided in analysis specifications. Further details are available at the URL below.
URL: http://www.amgen.com/datasharing

REFERENCES:
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com